CLINICAL TRIAL: NCT02586558
Title: Effect of Prebiotic on Colic and Crying and Fussing Behaviour in Infants CRI Study: Colic Relief Initiative Study
Brief Title: Effect of a Prebiotic on Colic and Crying and Fussing Behaviour in Infants
Acronym: CRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: McMaster University (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Principal Investigator, John Cairney, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCH-681
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Infant Formula (Active Comparator): Milk-based infant formula with prebiotics
  Interventions: Other: Experimental Infant formula
- Reference group (Placebo Comparator): Milk-based infant formula without prebiotics
  Interventions: Other: Reference group

INTERVENTIONS:
Other: Experimental Infant formula — Ready-to-feed infant formula to be fed ad libitum
  Arms: Experimental Infant Formula
Other: Reference group — Ready-to-feed infant formula to be fed ad libitum
  Arms: Reference group

SUMMARY:
Colic, or inconsolable crying and fussing, affects around 20% of babies who are 3 months of age or younger. To date, there are no known treatments that have been found to help reduce colic and its symptoms in babies. The investigators would like to see whether a baby formula that contains a prebiotic will lead to the same improvements in babies with colic. The investigators will test this by giving some babies a formula with the prebiotic and other babies a placebo formula.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term infant from a singleton birth (=>37 weeks gestational age); formula fed; primary caregiver able to read and write in English; current colicky behaviour

Exclusion Criteria:

* Infants with known genetic syndromes; birth weight (<2500g); use of proton pump inhibitors; use of antibiotics in previous week; use of nutritional colic remedies; use of probiotics; maternal medical history of diabetes (excluding gestational diabetes), tuberculosis, or any perinatal infection while pregnant with child enrolled in study; presence of blood in infant stool sample; possible cow milk protein allergy

Ages: 2 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Infant crying and fussing behaviour | 6 weeks
  As assessed by the Barr Baby Behavior Diary

SECONDARY OUTCOMES:
Infant crying and fussing behaviour | 6 weeks
  As assessed by actigraphy and accelerometry
Stool Microbiota | 6 weeks
Stool calprotectin | 6 weeks
Parent satisfaction | 6 weeks
  As assessed by parent survey
Infant behaviour | 6 weeks
  As assessed by parent survey
Infant feeding patterns | 6 weeks
  As assessed by parent survey
Infant stool patterns | 6 weeks
  As assessed by parent survey
Postnatal depression | 6 weeks
  As assessed by parent survey

CONTACTS AND LOCATIONS:
Overall Officials: John Cairney, PhD, Principal Investigator — McMaster University
Locations (1):
- David Braley Health Sciences Centre, Hamilton, Ontario, Canada